CLINICAL TRIAL: NCT03117881
Title: Comparative Effectiveness Trial Between a Clinic- and Home-Based Complementary and Alternative Medicine Telerehabilitation Intervention for Adults With Multiple Sclerosis (MS)
Brief Title: Tele-Exercise and Multiple Sclerosis
Acronym: TEAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Alabama Neurology Associates, PC (Other); Lakeshore Foundation (Other)
Responsible Party: Principal Investigator, James Rimmer, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F161017003; MS-1511-33653 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2017-04-05; First posted 2017-04-18 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Yoga; Pilates; Telerehabilitation; Physical activity
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DirectCAM (Experimental): The DirectCAM arm receives the intervention content via therapists at participating clinics.
  Interventions: Behavioral: DirectCAM
- TeleCAM (Experimental): The TeleCAM arm receives the intervention content at home using pre-loaded tablets and Interactive Voice Response (IVR) system technology.
  Interventions: Behavioral: TeleCAM
- rDirectCAM (Experimental): The rDirectCAM arm is being implemented in response to Covid-19. The rDirectCAM arm receives the intervention content delivered remotely in real-time by therapists via videoconferencing technology.
  Interventions: Behavioral: rDirectCAM

INTERVENTIONS:
Behavioral: DirectCAM — The intervention consists of a 60-minute Complementary Alternative Medicine (CAM) program that includes yoga, Pilates and dual-functioning exercises, which is delivered 2 times per week for the first 8 weeks and 1 time per week for the following 4 weeks at a clinic with a therapist. At the end of week 12, participants will be asked to continue the program in their home for up to 1 year post-intervention using handouts.
  Arms: DirectCAM
Behavioral: TeleCAM — The intervention consists of a 60-minute Complementary Alternative Medicine (CAM) program that includes yoga, Pilates and dual-functioning exercises, which is delivered 2 times per week for the first 8 weeks and 1 time per week for the following 4 weeks at home via videos. At the end of week 12, participants will be asked to continue the program in their home for up to 1 year post-intervention using the videos.
  Arms: TeleCAM
Behavioral: rDirectCAM — The intervention consists of a 60-minute Complementary Alternative Medicine (CAM) program that includes yoga, Pilates and dual-functioning exercises, which is delivered 2 times per week for the first 8 weeks and 1 time per week for the following 4 weeks by a therapist via videoconferencing technology. At the end of week 12, participants will be asked to continue the program in their home for up to 1 year post-intervention using handouts.
  Arms: rDirectCAM

SUMMARY:
The purpose of this study is to compare the effects of two delivery models of an evidence-based complementary alternative medicine (CAM) program that combines neurorehabilitative (functional) exercise, yoga, and Pilates for adults age 18-70 with multiple sclerosis (MS). CAM will be delivered as a 12-week program through two different delivery forms: On-site at a clinic (DirectCAM) and telerehabilitation (TeleCAM). Participants will be randomly assigned to one of these two groups.

**On March 16th, 2020, the University of Alabama at Birmingham halted all onsite non-essential research in response to the Covid-19 pandemic. Since then, the study has begun to conduct all testing remotely through videoconferencing technology. In addition, another study group, remote DirectCAM (rDirectCAM), has been incorporated into the study to continue the 12-week program delivery for newly recruited participants via videoconferencing technology.**

DETAILED DESCRIPTION:
There are few primary care and multiple sclerosis (MS) clinics that provide full exercise and rehabilitation services for patients with MS, especially in mostly rural, low-income areas such as Alabama, Mississippi, and Tennessee. Telerehabilitation, or the delivery of rehabilitation services over the telephone and/or the Internet, can help fill service gaps for underserved MS patient populations in this region. The proposed study will determine if our evidence-based rehabilitation and exercise program produces similar health outcomes when delivered in clinic or at home, using pre-loaded tablets and Interactive Voice Response (IVR) system technology among 759 participants with MS from 40 clinics across Alabama, Mississippi, and Tennessee.

**In response to the Covid-19 pandemic, the study aims to recruit 74 participants with MS into the rDirectCAM, where the 12-week program is delivered in real-time via videoconferencing technology. The rDirectCAM will determine if a telehealth rehabilitation program can have a similar effect as when the program is offered in person.**

The outcomes that we hope to achieve through the proposed rehabilitation and exercise program, referred to as complementary alternative medicine, are improved physical activity, decreased pain and fatigue, and quality of life. We also seek to improve attitudes and behaviors related to physical activity, such as outcome expectations for physical activity, social support from family and friends for physical activity, self-eﬃcacy (i.e., confidence in one's ability to be active), and self-regulation (i.e., setting exercise goals). We will examine the variation in outcomes by patient characteristics such as age and severity of disability to determine for whom the intervention is effective.

This project is important to patients with MS because it seeks to reduce their barriers to receiving exercise treatment and increase the convenience and appeal of such programs through technology. Furthermore, findings and resources from this study will be quickly provided to MS patients and clinicians across the United States (e.g., via training webinars through our National Center on Health, Physical Activity, and Disability [NCHPAD]) and thereby improve the quality and reach of exercise treatment for patients with MS.

The patient and stakeholder partners include MS patients, caretakers, and clinicians, who have been actively guiding the development of this project. In stakeholder meetings, members have provided insight into exercise treatment needs and preferences (e.g., individually tailored approaches that account for varying levels of mobility); outcomes of interest to the patient population (e.g., pain, fatigue, quality of life); and strategies for engaging/motivating participants with MS who may be discouraged and experiencing fatigue and pain (e.g., IVR calls and feedback). Moreover, their ongoing program satisfaction feedback will be important to our recruitment and retention success. Finally, the stakeholders will help make this project successful by continuing to emphasize the importance of long-term gains in health outcomes and promote (through NCHPAD) the sustainability of the program.

ELIGIBILITY:
Inclusion Criteria:

* Physician permission to participate in the study
* Mild to moderate disability (i.e., ambulate with/without assistive device, Patient-Determined Disease Steps [PDDS] 0 - 7
* Able to use arms/legs for exercise

Exclusion Criteria:

* Significant visual acuity that prevents seeing a tablet screen to follow home exercise program
* Cardiovascular disease event within the last six months, several pulmonary disease, and/or renal failure
* Active pressure ulcers
* Currently pregnant
* Within 30 days of receiving a rehabilitation program
* Already meeting physical activity guidelines (GLTEQ > 24)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 911 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Upstream Rehabilitation Inc., Athens, Alabama
  - Upstream Rehabilitation Inc., Bessemer, Alabama
  - Tanner Foundation, Birmingham, Alabama
  - Upstream Rehabilitation Inc., Calera, Alabama
  - Upstream Rehabilitation Inc., Cullman, Alabama
  - Southeast Alabama Medical Center Rehabilitation Services, Dothan, Alabama
  - Gulf Coast Therapy, Fairhope, Alabama
  - Gulf Coast Therapy, Foley, Alabama
  - Encore Rehabilitation, Fort Payne, Alabama
  - Upstream Rehabilitation Inc., Gadsden, Alabama
  - Therapy Achievements, Huntsville, Alabama
  - Upstream Rehabilitation Inc., Jacksonville, Alabama
  - Upstream Rehabilitation Inc., Jasper, Alabama
  - Gulf Coast Therapy, Mobile, Alabama
  - Montgomery East Physical Therapy, Montgomery, Alabama
  - Upstream Rehabilitation Inc., Muscle Shoals, Alabama
  - Encore Rehabilitation, Phenix City, Alabama
  - Upstream Rehabilitation Inc., Tuscaloosa, Alabama
  - Cornerstone Rehabilitation, Batesville, Mississippi
  - Upstream Rehabilitation Inc., Byram, Mississippi
  - Upstream Rehabilitation Inc., Canton, Mississippi
  - Upstream Rehabilitation Inc., Columbus, Mississippi
  - Upstrem Rehabilitation, Forest, Mississippi
  - Upstream Rehabilitation Inc., Fulton, Mississippi
  - River City Rehabilitation, Greenville, Mississippi
  - Encore Rehabilitation, Grenada, Mississippi
  - Upstream Rehabilitation Inc., Hattiesburg, Mississippi
  - Methodist Rehabilitation Center, Jackson, Mississippi
  - Encore Rehabilitation, Ocean Springs, Mississippi
  - North Sunflower Medical Center, Ruleville, Mississippi
  - Cornerstone Rehabilitation, Southaven, Mississippi
  - Upstream Rehabilitation Inc., Starkville, Mississippi
  - Upstream Rehabilitation Inc., Tupelo, Mississippi
  - Cornerstone Rehabilitation, Water Valley, Mississippi
  - Upstream Rehabilitation Inc., Bristol, Tennessee
  - Upstream Rehabilitation Inc., Cool Springs, Tennessee
  - Upstream Rehabilitation Inc., Gordonsville, Tennessee
  - Upstream Rehabilitation Inc., Knoxville, Tennessee
  - Upstream Rehabilitation Inc., Newport, Tennessee
  - Upstream Rehabilitation Inc., Winchester, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tracy TF, Young HJ, Lai B, Layton B, Stokes D, Fry M, Mehta T, Riser ES, Rimmer J. Supporting successful recruitment in a randomized control trial comparing clinic and home-based exercise among adults with multiple sclerosis. Res Involv Engagem. 2022 Jul 29;8(1):35. doi: 10.1186/s40900-022-00366-6. PMID 35906699
- [Derived] Lai B, Chiu CY, Pounds E, Tracy T, Mehta T, Young HJ, Riser E, Rimmer J. COVID-19 Modifications for Remote Teleassessment and Teletraining of a Complementary Alternative Medicine Intervention for People With Multiple Sclerosis: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jul 3;9(7):e18415. doi: 10.2196/18415. PMID 32540838
- [Derived] Rimmer JH, Thirumalai M, Young HJ, Pekmezi D, Tracy T, Riser E, Mehta T. Rationale and design of the tele-exercise and multiple sclerosis (TEAMS) study: A comparative effectiveness trial between a clinic- and home-based telerehabilitation intervention for adults with multiple sclerosis (MS) living in the deep south. Contemp Clin Trials. 2018 Aug;71:186-193. doi: 10.1016/j.cct.2018.05.016. Epub 2018 May 30. PMID 29859267

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Started | 425 | 412 | 74
Completed | 382 | 377 | 74
Not Completed | 43 | 35 | 0
Not completed — Withdrawal by Subject | 21 | 10 | 0
Not completed — Lost to Follow-up | 22 | 25 | 0
Period: Post-Intervention Follow-Up (3 Months)
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Started | 382 | 377 | 74
Completed | 289 | 296 | 67
Not Completed | 93 | 81 | 7
Not completed — Withdrawal by Subject | 26 | 21 | 1
Not completed — Lost to Follow-up | 34 | 38 | 4
Not completed — Did not complete test | 33 | 22 | 2
Period: 6-Month Follow-Up
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Started | 344 | 318 | 69
Completed | 269 | 277 | 60
Not Completed | 75 | 41 | 9
Not completed — Withdrawal by Subject | 4 | 8 | 0
Not completed — Lost to Follow-up | 18 | 8 | 2
Not completed — Did not complete test | 53 | 25 | 7
Period: 12-Month Follow-Up
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Started | 322 | 302 | 0
Completed | 261 | 278 | 0
Not Completed | 61 | 24 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0
Not completed — Lost to Follow-up | 18 | 22 | 0
Not completed — Did not complete test | 40 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DirectCAM | TeleCAM | rDirectCAM | Total
Number analyzed (Participants) | 382 | 377 | 74 | 833
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.3) | 50.0 (11.0) | 49.3 (11.7) | 50.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341 | 335 | 62 | 738
  Male | 41 | 42 | 12 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 94 | 86 | 20 | 200
  White | 278 | 278 | 53 | 609
  More than one race | 1 | 6 | 0 | 7
  Unknown or Not Reported | 7 | 6 | 1 | 14
Region of Enrollment [Number; unit: participants]
  United States | 382 | 377 | 74 | 833
Pain measured by 36-Item Short Form Survey (SF-36) Pain domain [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 382 | 377 | 68 | 827
    (all) | 56.84 (23.88) | 58.64 (24.62) | 60.70 (25.85) | 57.98 (24.38)
Fatigue measured by Modified Fatigue impact Scale [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 375 | 368 | 68 | 811
    (all) | 43.64 (16.80) | 42.84 (16.98) | 40.19 (19.50) | 42.99 (17.12)
Quality of life measured by 36-Item Short Form Survey (SF-36) physical component score [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 355 | 350 | 68 | 773
    (all) | 35.03 (11.30) | 35.80 (11.21) | 39.30 (11.43) | 35.75 (11.32)
Quality of life measured by 36-Item Short Form Survey (SF-36) mental component score [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 355 | 350 | 68 | 773
    (all) | 42.77 (14.78) | 43.05 (14.67) | 41.71 (14.94) | 42.80 (14.73)
Physical activity measured by Godin Leisure Time Exercise Score [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 319 | 330 | 68 | 717
    (all) | 14.16 (16.56) | 17.72 (55.70) | 3.16 (3.73) | 14.75 (39.57)
Balance measured by Berg Balance Scale [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 382 | 375 | 44 | 801
    (all) | 44.16 (14.27) | 47.37 (12.18) | 52.07 (7.26) | 46.10 (13.18)
Balance measured by Five Times Sit to Stand [Mean (Standard Deviation); unit: seconds] — Population: The number is less than the total because of missing values in the data.
  seconds
    number analyzed (Participants) | 363 | 367 | 48 | 778
    (all) | 19.55 (12.48) | 17.88 (9.25) | 15.79 (6.68) | 18.53 (10.80)
Endurance measured by Six Minute Walk Test [Mean (Standard Deviation); unit: meters] — Population: The number is less than the total because of missing values in the data.
  meters
    number analyzed (Participants) | 358 | 359 | 0 | 717
    (all) | 296.98 (127.19) | 317.74 (124.48) |  | 307.38 (126.18)
Gait measured by Timed Up and Go [Mean (Standard Deviation); unit: seconds] — Population: The number is less than the total because of missing values in the data.
  seconds
    number analyzed (Participants) | 371 | 370 | 44 | 785
    (all) | 16.89 (25.06) | 14.50 (21.05) | 9.82 (5.52) | 15.37 (22.58)
Gait measured by Timed 25-Foot Walk Test [Mean (Standard Deviation); unit: seconds] — Population: The number is less than the total because of missing values in the data.
  seconds
    number analyzed (Participants) | 366 | 363 | 0 | 729
    (all) | 11.72 (27.53) | 8.38 (9.62) |  | 10.06 (20.70)
Grip strength measured by hand dynamometer [Mean (Standard Deviation); unit: pounds] — Population: The number is less than the total because of missing values in the data.
  pounds
    number analyzed (Participants) | 377 | 365 | 49 | 791
    (all) | 50.86 (20.58) | 51.41 (19.45) | 49.13 (19.97) | 51.01 (20.01)
Outcome Expectations for Exercise measured by Multidimensional Outcome Expectations for Exercise [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 376 | 377 | 68 | 821
    (all) | 60.16 (7.39) | 60.51 (7.54) | 59.22 (6.48) | 60.25 (7.39)
Exercise Self Efficacy measured by Exercise Self-Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 377 | 376 | 68 | 821
    (all) | 80.90 (16.71) | 91.14 (14.27) | 87.56 (18.08) | 90.28 (15.78)
Social Support for Exercise measured by Social Provisions Scale [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 377 | 374 | 68 | 819
    (all) | 12.39 (2.12) | 12.27 (2.06) | 15.65 (1.93) | 12.61 (2.27)
Exercise Self Regulation measured by Exercise Goal-Setting Scale [Mean (Standard Deviation); unit: units on a scale] — Population: The number is less than the total because of missing values in the data.
  units on a scale
    number analyzed (Participants) | 380 | 362 | 68 | 810
    (all) | 23.28 (10.06) | 23.47 (9.45) | 20.29 (9.44) | 23.12 (9.76)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain
Description: Pain was measured by 36-Item Short Form Survey (SF-36). The score ranges from 0 to 100, with a higher score indicating less pain.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for rDirectCAM reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 382 | 377 | 68
score on a scale | 1.64 [-0.60 to 3.88] | 1.53 [-0.72 to 3.78] | -2.12 [-7.40 to 3.15]

2. Primary Outcome: Change in Fatigue
Description: Fatigue was measured by Modified Fatigue Impact Scale (MFIS). The total score range is 0 to 84, with a higher score indicating more fatigue.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 375 | 368 | 68
score on a scale | -2.57 [-3.90 to -1.24] | -3.58 [-4.92 to -2.23] | -1.36 [-4.49 to 1.77]

3. Primary Outcome: Change in Quality of Life (Physical Component)
Description: The physical component of quality of life was measured by the 36-Item Short Form Survey (SF-36) Physical Component score. The score ranges from 0 to 100, with higher scores indicating better quality of life in the physical component.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 355 | 350 | 68
score on a scale | 1.34 [0.36 to 2.86] | 1.86 [0.91 to 2.86] | 0.70 [-1.44 to 2.83]

4. Primary Outcome: Change in Quality of Life (Mental Component)
Description: The mental component of quality of life was measured by the 36-Item Short Form Survey (SF-36) Mental Component score. The score ranges from 0 to 100, with higher scores indicating better quality of life in the mental component.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 355 | 350 | 68
score on a scale | 0.42 [-1.06 to 1.90] | 1.10 [-0.38 to 2.57] | -1.09 [-4.38 to 2.19]

5. Primary Outcome: Change in Physical Activity
Description: Measured by the Godin Leisure Time Exercise Questionnaire (GLTEQ). The score ranges from 0 to 119, with higher scores indicating more physical activity.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 319 | 330 | 68
score on a scale | 3.74 [-5.02 to 12.51] | 6.46 [-2.17 to 15.09] | 3.13 [-14.20 to 20.47]

6. Secondary Outcome: Change in Balance (Berg Balance Scale)
Description: Balance was measured using the Berg Balance Scale (BBS). The score ranges from 0 to 56, with a lower score indicating a higher risk of falling and a higher score indicating better functional mobility.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample sizes for TeleCAM and rDirectCAM reported in this outcome was lower than the sample sizes reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 382 | 375 | 44
score on a scale | 3.67 [3.14 to 4.21] | 1.56 [1.02 to 2.11] | 1.93 [000 to 3.86]

7. Secondary Outcome: Change in Balance (Five Times Site to Stand)
Description: Balance was measured by the Five Times Site to Stand (FTSTS) test. Less time (in seconds) used to complete the FTSTS test indicates better balance.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 363 | 367 | 48
seconds | -3.33 [-4.48 to -2.17] | -2.28 [-3.43 to -1.12] | -2.45 [-6.64 to 1.74]

8. Secondary Outcome: Change in Endurance
Description: Endurance was measured using the 6-Minute Walk Test (6MWT). More distance traveled (meters) within the 6 minutes indicates better walking endurance.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample sizes for DirectCAM and TeleCAM reported in this outcome was lower than the sample sizes reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM.
Population: The Six-Minute Walk test was not assessed for participants in the rDirectCAM arm.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 358 | 359 | 0
meters | 28.30 [19.36 to 37.25] | 23.04 [14.10 to 31.99] |

9. Secondary Outcome: Change in Gait (Timed Up and Go)
Description: Gait was measured by the Timed Up and Go (TUG) test. Less time (in seconds) taken to complete the TUG test indicates better gait.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 371 | 370 | 44
seconds | -2.24 [-4.03 to -0.45] | -1.20 [-3.00 to 0.60] | -1.72 [-8.66 to 5.22]

10. Secondary Outcome: Change in Gait (Timed 25-Foot Walk)
Description: Gait was measured using the Timed 25-Foot Walk (T25FW) test. Less time taken to complete the T25FW test indicates better gait.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample sizes for DirectCAM and TeleCAM reported in this outcome was lower than the sample sizes reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM.
Population: The Time 25-foot Walk was not assessed among the rDirectCAM arm.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 366 | 363 | 0
seconds | -0.86 [-2.86 to 1.15] | 0.48 [-1.53 to 2.50] |

11. Secondary Outcome: Change in Grip Strength
Description: Grip strength was measured using a hand-held dynamometer. The higher score measured in pounds (lbs) indicates better grip strength.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: lbs
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 377 | 365 | 49
lbs | 3.11 [1.54 to 4.67] | 2.68 [1.10 to 4.26] | 4.35 [-1.11 to 9.81]

12. Other Pre Specified Outcome: Change in Outcome Expectations for Exercise
Description: Outcome expectations for exercise was measured by the Multidimensional Outcome Expectations for Exercise Scale (MOEES). The total score ranges from 15 to 75, with a higher score on the MOEES reflects greater positive expectations regarding the outcomes of exercise across the three domains (physical, social, and self-evaluative).
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample sizes for DirectCAM and rDirectCAM reported in this outcome was lower than the sample sizes reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 376 | 377 | 68
score on a scale | -1.00 [-1.91 to -0.10] | -0.21 [-1.12 to 0.70] | -0.48 [-2.51 to 1.56]

13. Other Pre Specified Outcome: Change in Exercise Self-Efficacy
Description: Exercise self-efficacy was measured by the Exercise Self-Efficacy Scale. The total score ranges from 0 to 100, with higher scores indicate better exercise self-efficacy.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 377 | 376 | 68
score on a scale | -27.0 [-30.24 to -23.70] | -26.98 [-30.25 to -23.69] | -4.41 [-11.35 to 2.54]

14. Other Pre Specified Outcome: Change in Social Support for Exercise
Description: Social support for exercise was measured by the Social Provisions Scale. The score ranges from 24 (1 point for each item) to 96 (4 points for each item), with higher scores indicate higher perceived social support and lower scores suggest lower perceived social support.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 377 | 374 | 68
score on a scale | 1.24 [0.94 to 1.54] | 1.38 [1.08 to 1.69] | 0.33 [-0.32 to 0.98]

15. Other Pre Specified Outcome: Change in Exercise Self-Regulation
Description: Exercise self-regulation was measured by the Exercise Goal-Setting Scale. The total score ranges from 10 to 50, with a higher score indicates better or more effective goal-setting behaviors in relation to exercise.
  The change was estimated at Month 12 compared to baseline for DirectCAM and TeleCAM, and at Month 3 compared to baseline for rDirectCAM. The mean difference and 95% confidence interval of this outcome were reported based on mixed models analyzed using intent-to-treat approach, including all available baseline data for the outcome. Please note that while some participants completed baseline, not all outcome measures were completed. As a result, the sample size for each arm reported in this outcome was lower than the sample size reported in the Participant Flow Overview section.
Time Frame: 48 weeks for DirectCAM and TeleCAM and 12 weeks for rDirectCAM.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
Number analyzed (Participants) | 380 | 376 | 68
score on a scale | 0.46 [-0.57 to 1.49] | 3.63 [2.60 to 4.67] | 3.71 [1.13 to 6.28]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | DirectCAM | TeleCAM | rDirectCAM
All-Cause Mortality (participants affected / at risk) | 0/425 | 0/412 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/425 | 2/412 | 0/74
Other Adverse Events (participants affected / at risk) | 0/425 | 0/412 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DirectCAM (N=425) | TeleCAM (N=412) | rDirectCAM (N=74)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Participant was hospitalized due to a seizure and later diagnosed with urinary tract infection. Participant had MRI and CT and was prescribed antibiotic and Keppra. The study follow-up test was rescheduled and participant later completed the test.
Hospitalized due to Covid-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Participant was hospitalized due to Covid-19 and bilateral pneumonia. Participant was on IV for hydration and antibiotics for pneumonia. The study follow-up test was rescheduled and participant later completed the test.

LIMITATIONS AND CAVEATS:
Our study had some limitations, which include: 1) limitations in reimbursement for onsite clinic services; 2) apprehension and competency in using technology; 3) difficulty in following participants residing in low resource communities over time; 4) challenge in identifying rural clinic sites, resulting in less than 10% of our participants from rural areas; 5) much higher percentage of female participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03117881/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03117881/ICF_001.pdf